CLINICAL TRIAL: NCT03718793
Title: Small Airway Inflammation and Dysfunction in Different Asthma Phenotypes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Lauri Lehtimäki, Associate professor, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R17004
Record Dates: First submitted 2018-10-11; First posted 2018-10-24 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects with asthma (Experimental): In addition to normal diagnostic work out we will measure small airway inflammation based on peripheral exhaled nitric oxide and assess small airway dysfunction using impulse oscillometry. In addition, inflammatory markers in peripheral blood and genotype will be assessed.
  Interventions: Diagnostic Test: Peripheral exhaled nitric oxide

INTERVENTIONS:
Diagnostic Test: Peripheral exhaled nitric oxide — Small airway inflammation and dysfunction will be measured using the above mentioned tests.
  Other Names: Impulse oscillometry; ECP/B-eos ratio

SUMMARY:
Small airway inflammation and dysfunction will be measured in 40 children and 40 adults with asthma before and after 8 weeks of treatment with inhaled budesonide. The same measurements will be conducted once in 80 age and sex matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of asthma and objective evidence of variable or reversible airway obstruction according to at least one of the following criteria
* significant response to bronchodilator (in subjects 7 years or older: FEV1 (forced expiratory volume in 1st second) or FVC (forced vital capacity) increases at least 12 % and 200 ml; in 4-6 years old subjects R5 decreases at least 40 %)
* in at least 12 years old subjects significant diurnal variation (at least 20 % and 60 l/min on at least three days) or significant response to bronchodilator ( at least 15 % and 60 l/min on at least three occasions) in PEF (peak expiratory flow) during a two-week monitoring
* significant airway hyperreactivity (PD20 FEV1 of methacholine less than 600 µg in at least 16 years old subjects, FEV1 decreases at least 15 % in exercise test in 7-15 years old, or R5 increases at least 40 % during free-running test in 4-6 years old subjects)

Exclusion Criteria:

* current smoking
* regular anti-inflammatory asthma medication (will be paused for at least 4 weeks before enrollment)
* other chronic pulmonary disease
* other diseases that in the opinion of the treating physician prevents participation

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of small airway inflammation (measured by peripheral NO output) in untreated asthma | Baseline
  Change in peripheral NO output
Prevalence of small airway dysfunction (measured by peripheral airway resistance) in untreated asthma | Baseline
  Change in peripheral airway resistance

SECONDARY OUTCOMES:
Difference in Eosinophil Cationic Protein (ECP)/B-Eos ratio between asthmatics and controls | Baseline
  ECP/B-Eos ratio will calculated by dividing serum level of ECP by peripheral blood eosinophil count.
Correlation between ECP/B-Eos ratio and peripheral NO output in untreated asthma | Baseline
  ECP/B-Eos ratio will be calculated as above. Peripheral exhaled NO output will be calculated based on exhaled NO measurement at multiple flow rates.
Correlation between ECP/B-Eos ratio and peripheral airway resistance in untreated asthma | Baseline
  ECP/B-Eos ratio will be calculated as above. Peripheral airway resistance will be calculated as R5-R20 based on impulse oscillometry.

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Lehtimäki, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Allergy Centre, Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No